CLINICAL TRIAL: NCT03792607
Title: Perturbation of Interactome Through Micro-RNA And Methylome Analyses In Diabetes Endophenotypes: the PIRAMIDE Study Design
Brief Title: Network-based Approach in Type 2 Diabetes and Its Cardiovascular Risk
Acronym: PIRAMIDE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Giuditta Benincasa (Other)
Responsible Party: Sponsor-Investigator, Giuditta Benincasa, Principal Investigator GIUDITTA BENINCASA, University of Campania Luigi Vanvitelli
Organization: University of Campania Luigi Vanvitelli (Other)
Other Study IDs: RRC-2015-2360454
Record Dates: First submitted 2018-12-21; First posted 2019-01-03 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes Mellitus; Cardiovascular Diseases
Keywords: Network medicine; Epigenetics; Diabetes; Cardiovascular risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood CD4+ T cells and CD8+ T cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
PIRAMIDE study design will test the hypothesis that simultaneous interactions between DNA methylation and microRNAs may hit T2D candidate genes and predict the development of T2D-related cardiovascular complications.

ELIGIBILITY:
Exclusion Criteria:

* Clinical Diagnosis of Type 2 Diabetes. In according to current guidelines, diabetes is diagnosed by evidence of impairing fast glucose (IFG) > 7.0 mmol/L (>125 mg/dl), post prandial glycemia > 11.1 mmol/L (>200 mg/dl), and evidence of glycated hemoglobin (HbA1c) > 6.6%. Clinical and demographic characteristics of study population will be avaiable from datasets generated by physicians.
* Clinical Diagnosis of macrovascular dysfunction.

Exclusion Criteria:

• Patients with known history of cancer, malignancy disorders, active infections, and chronic or immune-mediated diseases.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will enroll 35 men and women 50 years or older with diagnosis of T2D and 35 sex and age-matched controls. Population study will be recruited at the Department of Medical, Surgical, Neurological, Metabolic and Geriatric Sciences of University della Campania "Luigi Vanvitelli".
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-01-14 (Estimated); Study Completion 2020-06-14 (Estimated)

PRIMARY OUTCOMES:
DNA methylation status both of CD4+ and CD8+ cells | 3 Months
  Using Methylation 27K BeadChip platform based on Bisulfite conversion technology, DNA methylation profile of 35 preselected T2D patients will be measured both in CD4+ and CD8+ cells collected from peripheral blood respect with controls.
Bioinformatics analysis to predict putative novel T2D candidate genes | 6 Months
  The network-based algorithm "Weighted Human DNA methylation PPI network (WMPN)" will be applied to methylome data in order to obtain a disease module containing the crucial differentially methylated genes both in CD4+ and CD8+ cells from T2D patients and controls.
RNA sequencing analysis both in CD4+ and CD8+ cells | 3 Months
  RNA sequencing analysis by using Illumina HiSeq2000 Next Generatin Sequencing (NGS) platform will be performed for identifying differentially expressed micro-RNA and mRNA target both in CD4+ and CD8+ cells isolated from T2D patients and controls .

SECONDARY OUTCOMES:
ROC curves to evaluate putative DNA methylation/microRNA interactions as prognostic biomarkers of cardiovascular dysfunction in T2D patients | 12 Months
  The ROC curves will be used to correlation putative epigenetics interactions (DNA methylation and microRNA) with the presence or absence of T2D-related cardiovascular dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Giuditta Benincasa, MSc, Principal Investigator — Clinical Department of Internal Medicine and Specialistics
Locations (1):
- Università della Campania Luigi Vanvitelli, Naples, Italy

REFERENCES:
- [Derived] Benincasa G, Franzese M, Schiano C, Marfella R, Miceli M, Infante T, Sardu C, Zanfardino M, Affinito O, Mansueto G, Sommese L, Nicoletti GF, Salvatore M, Paolisso G, Napoli C. DNA methylation profiling of CD04+/CD08+ T cells reveals pathogenic mechanisms in increasing hyperglycemia: PIRAMIDE pilot study. Ann Med Surg (Lond). 2020 Oct 20;60:218-226. doi: 10.1016/j.amsu.2020.10.016. eCollection 2020 Dec. PMID 33194177